CLINICAL TRIAL: NCT04405115
Title: Improving Survivorship Care for Older Adults After Chemotherapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019028
Record Dates: First submitted 2020-03-18; First posted 2020-05-28 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Survivorship
Keywords: survivorship care; Chemo; chemotherapy; older; survivor
MeSH Terms: interventions — Geriatric Assessment

STUDY DESIGN:
Intervention Model Description: 2 arms; 1:1 randomization;
  Standard of care (control group) will receive routine care only and will not be scheduled for a Comprehensive Geriatric Assessments visit.
  Comprehensive geriatric assessment ( intervention group) will be scheduled for a Comprehensive Geriatric Assessment visit that will take place with a geriatric nurse practitioner of a physician as soon as possible following enrollment and randomization (preferably within 2 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention arm (No Intervention): routine care only; will not be scheduled for comprehensive geriatric assessment
- Active comparator arm (Active Comparator): those that will be scheduled for comprehensive geriatric assessment with a geriatric nurse practitioner or physician
  Interventions: Behavioral: Geriatric Assessment

INTERVENTIONS:
Behavioral: Geriatric Assessment — Geriatric Assessment Visit
  Arms: Active comparator arm

SUMMARY:
The researchers want to find out if older adults receiving a survivorship care plan followed by a geriatric assessment visit improves quality of life and satisfaction with care compared to receiving only a survivorship care plan for older adults who have completed chemotherapy for cancer treatment.

DETAILED DESCRIPTION:
This study is a pilot randomized trial to examine whether a geriatric assessment-enhanced survivorship care plan improves satisfaction, knowledge and health-related quality of life compared to standard survivorship care plans among older adults who have completed curative chemotherapy for cancer. The investigator's hypothesis is that older adults who receive a geriatric assessment-enhanced survivorship care plan will report improved satisfaction with care, health-related quality of life, and knowledge and preparedness for survivorship care needs.

ELIGIBILITY:
Inclusion Criteria:

1. age 65 years and above and
2. Have diagnosis of cancer and have completed chemotherapy with curative (not palliative) intent and
3. have been scheduled to receive a survivorship care plan from an oncology navigator.

Exclusion Criteria:

1. advanced dementia or serious cognitive impairment that would impede ability to participate in the interview
2. nursing home resident.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-02-16 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Study retention rate | 4-6 months
  Feasibility of the study will be assessed by study retention rate which is defined as proportion of enrolled participants who remain enrolled until study completion.
Number of months needed for completion of trial enrollment | 4-6 months
Acceptability of the study: survey | 4-6 months
  Assess acceptability via a short survey administered to participating oncology nurse navigators and patients selected for the intervention group.

SECONDARY OUTCOMES:
Patient satisfaction assessment by PSCC (Patient Satisfaction with Cancer related Care) tool | 4-6 months
  PSCC items are rated on 5-point Likert scales: "1 = Strongly Agree", "2 = Agree", "3 = Neutral", "4 = Disagree", and "5 = Strongly Disagree". A lower PSCC total score indicates higher satisfaction level
Health related quality of life assessment by the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire EORTC QLQ-30 | 4-6 months
  The QLQ-C30 questionnaire is a specific questionnaire for cancer, it is composed of 30 questions or items that assess the quality of life in relation to physical, emotional, social aspects and in general the level of functionality of patients diagnosed with cancer. The QLQ-C30 questionnaire is assigned values between 1 and 4 (1: not at all, 2: a little, 3: a lot, 4: a lot) according to the patient's responses to the item, only in items 29 and 30 are assessed with score from 1 to 7 (1: bad, 7: excellent). The scores obtained are standardized and a score between 0 and 100 is obtained, 0 being the worst possible and 100 the best.
Health related quality of life assessment by QLQ14 | 4-6 months
  QLQ-ELD14 is a validated quality of life questionnaire for cancer patients aged ⩾70 years and it is used in conjunction with EORTC QLQ-30.QLQ-ELD14 comprises five scales (mobility, worries about others, future worries, maintaining purpose and burden of illness) and two single items (joint stiffness and family support)
Self rated patient knowledge and preparedness measured by PLANS assessment tool (Preparing for Life as a New Survivor) | 4-6 months
  Preparing for Life as a New Survivor (PLANS) survey is utilized to evaluate survivor satisfaction with 1) own knowledge of diagnosis, treatment, and side effects, and 2) communication with the cancer team regarding diagnosis, treatment, and side effects.PLANS questions assess the level of agreement with statements regarding satisfaction with a 4-point scale (strongly disagree, somewhat disagree, somewhat agree, strongly agree) for each statement.

CONTACTS AND LOCATIONS:
Overall Officials: Haifaa Abdulhaq, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Community Cancer Institute, Clovis, California, United States

IPD SHARING:
Plan to Share IPD: No